CLINICAL TRIAL: NCT03057821
Title: Does Hydrogen Peroxide Skin Preparation Reduce Propionibacterium Acnes in Shoulder Arthroplasty?
Brief Title: Propionibacterium Acnes in Shoulder Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Peter Chalmers, Principle Investigator, University of Utah
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 96964
Record Dates: First submitted 2017-02-14; First posted 2017-02-20 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2019-08

CONDITIONS: Propionibacterium Acnes
Keywords: hydrogen peroxide; Propionibacterium Acnes; shoulder arthroplasty
MeSH Terms: interventions — Hydrogen Peroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will not receive any hydrogen peroxide skin preparation
- Treatment (Experimental): The treatment group will also undergo skin preparation with 3% hydrogen peroxide.
  Interventions: Other: 3% hydrogen peroxide

INTERVENTIONS:
Other: 3% hydrogen peroxide — The treatment group will also undergo skin preparation with 3% hydrogen peroxide.
  Arms: Treatment

SUMMARY:
The investigator's plan to determine whether pre-operative skin preparation with hydrogen peroxide alters rates of P acnes culture positivity. They hypothesize that pre-operative skin preparation with hydrogen peroxide will reduce rates of P acnes culture positivity.

DETAILED DESCRIPTION:
Over half of all post-operative infections after shoulder arthroplasty are due to Propionibacterium acnes. Even in apparently "aseptic" revisions, nearly all cultures taken at the time of revision surgery are positive for P acnes, and thus low-grade infection with this bacteria may be a more common cause of failure than previously suspected. Current antibiotic prophylaxis methods are ineffective against P acnes. Despite intravenous cefazolin, P acnes can be cultured from the glenohumeral joint in 42% of patients undergoing primary total shoulder arthroplasty. Despite skin preparation with chlorhexidine, P acnes can be cultured from 73% of portal sites in arthroscopy. P acnes is further insensitive to alcohol. Dermatologists have long been treating P acnes as it is a primary cause of acne vulgaris. One of the most popular and effective treatments for acne vulgaris is topical benzoyl peroxide. A prior prospective clinical trial demonstrated that adding topical 5% benzoyl peroxide 48 hours prior to surgery reduced P acnes culture positivity to 6%. The downside of this treatment is that it must be applied by the patient, at home, for 48 hours prior to surgery. An additional downside is that benzoyl peroxide is a skin irritant that not all patients tolerate.

In aqueous environments, benzoyl peroxide rapidly decomposes into benzoic acid and hydrogen peroxide. Benzoic acid is a skin irritant and hydrogen peroxide is the active ingredient. Benzoyl peroxide is used instead of hydrogen peroxide because hydrogen peroxide breaks down into water and oxygen when exposed to light. Recently, stabilized forms of hydrogen peroxide have been developed and have been demonstrated to be equally effective to benzoyl peroxide in the treatment of acne vulgaris. One potential reason for hydrogen peroxide's efficacy against P acnes is that it is absorbed into the skin, addressing P acnes residing in sebaceous glands. To date, no studies have examined whether the addition of hydrogen peroxide to pre-operative skin preparation can reduce intra-operative P acnes culture positivity.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary shoulder arthroplasty

Exclusion Criteria:

* Patients with prior shoulder surgery.
* Patients with a symptomatic infection or history of infection, recent antibiotic use (within six weeks), or with clinical signs of infection such as an elevated ESR, CRP, positive aspiration cultures, or positive biopsy.
* Patients with a known hypersensitivity to hydrogen peroxide.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Positive P acnes culture | 2-weeks
  The primary outcome of the study will be P acnes culture positive results.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chalmers, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No